CLINICAL TRIAL: NCT01756235
Title: Physical ACtivity in patiEnts With Rheumatoid Arthritis Treated With Adalimumab in Routine Clinical Practice (PACE)
Brief Title: Physical Activity in Patients With Rheumatoid Arthritis Treated With Adalimumab in Routine Clinical Practice
Acronym: PACE
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-683
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Post-marketing observational study (PMOS) Protocol; Rheumatoid Arthritis; Physical Activity; Adalimumab; Humira®
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Rheumatoid Arthritis: Participants with rheumatoid arthritis treated with adalimumab in routine clinical practice.

SUMMARY:
The purpose of this study was to evaluate physical activity and its changes in participants with rheumatoid arthritis (RA) who were treated with adalimumab therapy in clinical practice.

DETAILED DESCRIPTION:
This post-marketing observational study was conducted in a multi-country, multi-center and single-arm format. Data were collected prospectively. Adult participants with diagnosis of RA who were assigned for treatment with adalimumab (Humira®) were eligible for participation. During this period four follow-up visits were planned for observation of the participant and documentation of data. Ideally, these visits should have been performed approximately 3 (V1), 6 (V2), 9 (V3) and 12 (V4) months after the baseline visit (V0).

ELIGIBILITY:
Inclusion Criteria:

* Had rheumatoid arthritis (RA) and is eligible to start and/or continue adalimumab therapy according to the local product label and prescription guidelines
* Had been started on adalimumab therapy no more than one (1) month prior to the study enrolment
* Had negative result of tuberculosis (TB) screening test or was receiving TB prophylaxis as per local guidelines
* Had provided written Authorization to the investigator to use and/or disclose personal and/or health data, or Informed Consent if requested by the Local Regulations

Exclusion Criteria:

* Was unable to walk either due to RA or a comorbid condition
* Was unable to perform basic self-care activities
* Had contraindications for treatment with adalimumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consisted of participants with rheumatoid arthritis (RA) who were treated with adalimumab as per locally approved label and prescription guidelines. The decision to be treated with adalimumab had to be independent from study inclusion.
Sampling Method: Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2012-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Smirnova, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 462 participants were enrolled: 460 were in the main analysis set (MAS) population; 2 were excluded from MAS, as adalimumab treatment was not documented within this study.
Period: Overall Study
Arm/Group | Participants With Rheumatoid Arthritis
Started | 462
Completed | 460
Not Completed | 2
Not completed — Adalimumab Treatment was not Documented | 2

BASELINE CHARACTERISTICS:
Population: Baseline analyses accounts for main analysis set (MAS) population (all participants who received at least 1 dose of study drug).
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 460
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.1)
Gender [Count of Participants; unit: Participants]
  Female | 378
  Male | 82

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Physical Activity Short Questionnaire to Assess Health-enhancing Physical Activity (SQUASH) Score
Description: The quantitative SQUASH score (scores range from 0 to 17010.000) is calculated as the sum of subscores that capture physical activity related to commuting activities (SQUASH-A), scores range from 0 to 4082.400, leisure time activities (SQUASH-B), scores range from 0 to 6123.600, household activities (SQUASH-C), scores range from 0 to 3402.000, and activity at work and school (SQUASH-D), scores range from 0 to 3402.000. The SQUASH score and its subscores has non-negative values. Higher values indicate a higher individual activity level.
Time Frame: Month 0 (baseline) and Month 12 (Last Observation Carried Forward (LOCF))
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 374
units on a scale | 870.0 (4517.8)

2. Secondary Outcome: Mean Change From Baseline in Total Physical Activity SQUASH Score
Description: as for outcome 1
Time Frame: Month 3, Month 6 and Month 9
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 356
units on a scale
  Month 3 (N=356) | 454.9 (3553.9)
  Month 6 (N=316) | 648.2 (3565.1)
  Month 9 (N=273) | 611.3 (4130.4)

3. Secondary Outcome: Mean Change From Baseline in SQUASH-A Scores
Description: SQUASH subscores capture physical activity. SQUASH-A subscore captures commuting activities, with scores ranging from 0 to 4082.400. The SQUASH subscores have non-negative values. Higher values indicate a higher individual activity level.
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 382
units on a scale
  Month 3 (N=368) | -91.6 (950.2)
  Month 6 (N=327) | -41.7 (957.4)
  Month 9 (N=281) | 3.5 (1052.4)
  Month 12 (N=265) | 10.4 (880.4)
  Month 12 LOCF (N=382) | -35.7 (1043.2)

4. Secondary Outcome: Mean Change From Baseline in SQUASH-B Scores
Description: SQUASH subscores capture physical activity. SQUASH-B subscore captures leisure time activities, with scores ranging from 0 to 6123.600. The SQUASH subscores have non-negative values. Higher values indicate a higher individual activity level.
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 375
units on a scale
  Month 3 (N=359) | 399.5 (2729.2)
  Month 6 (N=319) | 497.9 (2375)
  Month 9 (N=277) | 358.9 (2720.5)
  Month 12 (N=257) | 831.3 (3450.7)
  Month 12 LOCF (N=375) | 578.0 (3131.1)

5. Secondary Outcome: Mean Change From Baseline in SQUASH-C Scores
Description: SQUASH subscores capture physical activity. SQUASH-C subscore captures house-hold activities, with scores ranging from 0 to 3402.000. The SQUASH subscores have non-negative values. Higher values indicate a higher individual activity level.
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 379
units on a scale
  Month 3 (N=364) | 81.4 (1507.5)
  Month 6 (N=325) | 154.6 (1516.5)
  Month 9 (N=281) | 98.5 (1590.6)
  Month 12 (N=261) | 315.4 (1750)
  Month 12 LOCF (N=379) | 196.9 (1725.9)

6. Secondary Outcome: Mean Change From Baseline in SQUASH-D Scores
Description: SQUASH subscores capture physical activity. SQUASH-D subscore captures activity at work and school, with scores ranging from 0 to 3402.000. The SQUASH subscores have non-negative values. Higher values indicate a higher individual activity level.
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 382
units on a scale
  Month 3 (N=370) | 47.3 (823.2)
  Month 6 (N=330) | 27.2 (1102.3)
  Month 9 (N=284) | 170.2 (1263.7)
  Month 12 (N=266) | 136.2 (1733.3)
  Month 12 LOCF (N=382) | 96.4 (1536.8)

7. Secondary Outcome: Mean Change From Baseline in Disease Activity Index - 28 Joints (DAS28) Score
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Tender joint counts and swollen joint counts across 28 joints, C-reactive protein, and general health assessed via the visual analog scale (VAS) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 433
units on a scale
  Month 3 (N=431) | -2.4 (1.4)
  Month 6 (N=390) | -2.8 (1.5)
  Month 9 (N=362) | -3.0 (1.5)
  Month 12 (N=334) | -3.3 (1.5)
  Month 12 LOCF (N=433) | -2.9 (1.7)

8. Secondary Outcome: Percentage of Participants in Clinical Disease Remission (DAS28<2.6)
Description: Remission is defined as DAS28 of less than 2.6. The DAS28 is a validated index of rheumatoid arthritis disease activity. Tender joint counts and swollen joint counts across 28 joints, C-reactive protein (CRP), and general health assessed via the visual analog scale (VAS) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: Month 0, Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 459
percentage of participants
  Month 0 (N=459) | 0.7
  Month 3 (N=432) | 21.3
  Month 6 (N=390) | 30.3
  Month 9 (N=362) | 32.3
  Month 12 (N=334) | 37.4
  Month 12 LOCF (N=434) | 31.1

9. Secondary Outcome: Percentage of Participants With Low Disease Activity State (LDAS, DAS28<3.2)
Description: LDAS is defined as DAS28 of less than 3.2. The DAS28 is a validated index of rheumatoid arthritis disease activity. Tender joint counts and swollen joint counts across 28 joints, C-reactive protein (CRP), and general health assessed via the visual analog scale (VAS) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: Month 0, Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 459
percentage of participants
  Month 0 (N=459) | 1.3
  Month 3 (N=432) | 35.4
  Month 6 (N=390) | 46.4
  Month 9 (N=362) | 54.4
  Month 12 (N=334) | 66.2
  Month 12 LOCF (N=434) | 56.0

10. Secondary Outcome: Mean Change From Baseline in Total Physical Activity SQUASH Scores and Individual Physical Activity Categories' SQUASH Scores in Participants in Remission or LDAS
Description: This outcome analyses the quantitative SQUASH score and individual SQUASH scores by DAS28 categories. The quantitative SQUASH score (ranging from 0 to 17010.000) is calculated as the sum of subscores that capture physical activity related to commuting activities (SQUASH-A), leisure time activities (SQUASH-B), household activities (SQUASH-C) and activity at work and school (SQUASH-D). The SQUASH score and its subscores has non-negative values. Higher values indicate a higher individual activity level. DAS28 categories being assessed are remission (defined as DAS28 of less than 2.6) and LDAS (defined as DAS28 of less than 3.2).The DAS28 is a validated index of rheumatoid arthritis disease activity. Tender joint counts and swollen joint counts across 28 joints, C-reactive protein (CRP), and general health assessed via the visual analog scale (VAS) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10, with higher scores indicating higher disease activity.
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 214
units on a scale
  SQUASH (Month 3, N=198) | 473.3 (3417.8)
  SQUASH-A (Month 3, N=204) | -57.5 (609.4)
  SQUASH-B (Month 3, N=200) | 438.3 (2480.6)
  SQUASH-C (Month 3, N=200) | 87.0 (1617.6)
  SQUASH-D (Month 3, N=205) | -11.3 (762.1)
  SQUASH (Month 6, N=181) | 979.8 (3567.4)
  SQUASH-A (Month 6, N=187) | -23.2 (724.8)
  SQUASH-B (Month 6, N=183) | 761.0 (2383.3)
  SQUASH-C (Month 6, N=186) | 234.5 (1518.8)
  SQUASH-D (Month 6, N=189) | -8.6 (1142.7)
  SQUASH (Month 9, N=162) | 1209.8 (4126.9)
  SQUASH-A (Month 9, N=165) | 130.3 (874.0)
  SQUASH-B (Month 9, N=164) | 707.2 (2815.5)
  SQUASH-C (Month 9, N=165) | 255.9 (1713.8)
  SQUASH-D (Month 9, N=167) | 142.4 (1298.6)
  SQUASH (Month 12, N=167) | 1912.4 (4592.1)
  SQUASH-A (Month 12, N=171) | 80.7 (724.8)
  SQUASH-B (Month 12, N=167) | 1158.7 (3168.1)
  SQUASH-C (Month 12, N=169) | 470.7 (1898.4)
  SQUASH-D (Month 12, N=171) | 171.6 (1905.4)
  SQUASH (Month 12 LOCF, N=211) | 1494.8 (4513.8)
  SQUASH-A (Month 12 LOCF, N=214) | 53.4 (860.0)
  SQUASH-B (Month 12 LOCF, N=211) | 964.5 (3127.4)
  SQUASH-C (Month 12 LOCF, N=212) | 367.5 (1808.5)
  SQUASH-D (Month 12 LOCF, N=214) | 90.0 (1778.7)

11. Secondary Outcome: Mean Change From Baseline in Total Physical Activity SQUASH Scores and Individual Physical Activity Categories' SQUASH Scores in Participants Those Who Did Not Attain Remission or LDAS
Description: as for outcome 10
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 167
units on a scale
  SQUASH (Month 3, N=157) | 434.5 (3739.9)
  SQUASH-A (Month 3, N=163) | -134.8 (1255.7)
  SQUASH-B (Month 3, N=158) | 352.9 (3029.8)
  SQUASH-C (Month 3, N=163) | 75.1 (1370.3)
  SQUASH-D (Month 3, N=164) | 120.7 (893.0)
  SQUASH (Month 6, N=135) | 203.6 (3526.4)
  SQUASH-A (Month 6, N=140) | -66.5 (1202.3)
  SQUASH-B (Month 6, N=136) | 143.9 (2325.7)
  SQUASH-C (Month 6, N=139) | 47.6 (1512.2)
  SQUASH-D (Month 6, N=141) | 75.1 (1047.9)
  SQUASH (Month 9, N=111) | -262.1 (3995.1)
  SQUASH-A (Month 9, N=116) | -176.9 (1245.6)
  SQUASH-B (Month 9, N=113) | -146.6 (2503.3)
  SQUASH-C (Month 9, N=116) | -125.5 (1373.1)
  SQUASH-D (Month 9, N=117) | 209.8 (1216.5)
  SQUASH (Month 12, N=88) | 230.7 (4924.9)
  SQUASH-A (Month 12, N=94) | -117.6 (1102.0)
  SQUASH-B (Month 12, N=90) | 223.9 (3867.2)
  SQUASH-C (Month 12, N=92) | 30.1 (1403.4)
  SQUASH-D (Month 12, N=95) | 72.4 (1377.4)
  SQUASH (Month 12 LOCF, N=162) | 61.6 (4420.2)
  SQUASH-A (Month 12 LOCF, N=167) | -150.2 (1235.1)
  SQUASH-B (Month 12 LOCF, N=163) | 81.3 (3083.7)
  SQUASH-C (Month 12 LOCF, N=166) | -19.8 (1599.0)
  SQUASH-D (Month 12 LOCF, N=167) | 105.1 (1166.4)

12. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores range from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from baseline in the overall score indicates improvement.
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 396
units on a scale
  Month 3 (N=384) | -0.5 (0.6)
  Month 6 (N=345) | -0.7 (0.6)
  Month 9 (N=300) | -0.8 (0.6)
  Month 12 (N=284) | -0.9 (0.6)
  Month 12 LOCF (N=396) | -0.7 (0.7)

13. Secondary Outcome: Correlation Between Physical Activity (Total SQUASH Score and Individual Physical Activity Categories' SQUASH Scores) and DAS28 Scores
Description: The SQUASH and its subscores are instruments to measure the physical activity level, whereas the DAS28 measures disease activity. In order to evaluate the relationship between physical function and disease activity (as measured by the two scales), Pearson correlation coefficients were calculated for the SQUASH scores and the DAS28. A decrease in physical functioning is likely to be connected to stronger disease activity.
Time Frame: Month 0 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Number; unit: Correlation coeficient
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 432
Correlation coeficient
  SQUASH and DAS28 (Month 0, N=423) | -0.19
  SQUASH and DAS28 (Month 12 LOCF, N=386) | -0.21
  SQUASH-A and DAS28 (Month 0, N=431) | -0.06
  SQUASH-A and DAS28 (Month 12 LOCF, N=386) | -0.07
  SQUASH-B and DAS28 (Month 0, N=424) | -0.10
  SQUASH-B and DAS28 (Month 12 LOCF, N=386) | -0.17
  SQUASH-C and DAS28 (Month 0, N=429) | -0.19
  SQUASH-C and DAS28 (Month 12 LOCF, N=386) | -0.15
  SQUASH-D and DAS28 (Month 0, N=432) | -0.09
  SQUASH-D and DAS28 (Month 12 LOCF, N=386) | -0.08

14. Secondary Outcome: Correlation Between Physical Activity (Total SQUASH Score and Individual Physical Activity Categories' SQUASH Scores) and HAQ-DI Scores
Description: The SQUASH and its subscores are instruments to measure the physical activity level, whereas the HAQ-DI measures physical functioning. In order to evaluate the relationship between physical function and physical activity (as measured by the both scales), Pearson correlation coefficients were calculated for the SQUASH scores and the HAQ-DI. A decrease in physical functioning is likely to prohibit physical activity.
Time Frame: Month 0 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Number; unit: Correlation coeficient
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 430
Correlation coeficient
  SQUASH (Month 0, N=421) | -0.30
  SQUASH (Month 12 LOCF, N=385) | -0.22
  SQUASH-A (Month 0, N=429) | -0.16
  SQUASH-A (Month 12 LOCF, N=385) | -0.11
  SQUASH-B (Month 0, N=422) | -0.21
  SQUASH-B (Month 12 LOCF, N=385) | -0.19
  SQUASH-C (Month 0, N=427) | -0.20
  SQUASH-C (Month 12 LOCF, N=385) | -0.10
  SQUASH-D (Month 0, N=430) | -0.14
  SQUASH-D (Month 12 LOCF, N=385) | -0.10

15. Secondary Outcome: Mean Change From Baseline in Physical Activity (Total SQUASH Score and Individual Physical Activity Categories' SQUASH Scores) Influenced by Age Categories
Description: as for outcome 1
Time Frame: Month 0 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 382
units on a scale
  SQUASH (<65 years, N=297) | 1066.2 (4456.6)
  SQUASH (>=65 years, N=77) | 113.1 (4699.9)
  SQUASH A (<65 years, N=302) | -27.5 (1066.4)
  SQUASH A (>=65 years, N=80) | -66.7 (956.4)
  SQUASH B (<65 years, N=298) | 770.8 (2850.4)
  SQUASH B (>=65 years, N=77) | -167.8 (3972.9)
  SQUASH C (<65 years, N=300) | 189.5 (1779.6)
  SQUASH C (>=65 years, N=79) | 225.0 (1514.7)
  SQUASH D (<65 years, N=302) | 103.8 (1691.5)
  SQUASH D (>=65 years, N=80) | 68.3 (697.8)

16. Secondary Outcome: Mean Change From Baseline in Physical Activity (Total SQUASH Score and Individual Physical Activity Categories' SQUASH Scores) Influenced by Gender
Description: as for outcome 1
Time Frame: Month 0 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 382
units on a scale
  SQUASH (Male, N=70) | 1500.1 (5026.2)
  SQUASH (Female, N=304) | 724.9 (4388.7)
  SQUASH-A (Male, N=70) | -133.9 (1091.0)
  SQUASH-A (Female, N=312) | -13.7 (1032.8)
  SQUASH-B (Male, N=70) | 948.3 (3565.2)
  SQUASH-B (Female, N=305) | 493.0 (3022.8)
  SQUASH-C (Male, N=70) | 344.7 (1774.0)
  SQUASH-C (Female, N=309) | 163.4 (1716.0)
  SQUASH-D (Male, N=70) | 264.6 (1719.8)
  SQUASH-D (Female, N=312) | 58.6 (1493.0)

17. Secondary Outcome: Mean Change From Baseline in Physical Activity (Total SQUASH Score and Individual Physical Activity Categories' SQUASH Scores) Influenced by Education
Description: as for outcome 1
Time Frame: Month 0 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 382
units on a scale
  SQUASH (High School, N=195) | 831.7 (3946.1)
  SQUASH (Lower than High School, N=179) | 911.8 (5079.0)
  SQUASH-A (High School, N=198) | -45.2 (926.9)
  SQUASH-A (Lower than High School, N=184) | -25.5 (1158.0)
  SQUASH-B (High School, N=195) | 520.5 (2187.4)
  SQUASH-B (Lower than High School, N=180) | 640.4 (3910.3)
  SQUASH-C (High School, N=198) | 202.1 (1751.3)
  SQUASH-C (Lower than High School, N=181) | 191.2 (1702.5)
  SQUASH-D (High School, N=198) | 131.4 (1644.3)
  SQUASH-D (Lower than High School, N=184) | 58.7 (1415.5)

18. Secondary Outcome: Mean Change From Baseline in Physical Activity (Total SQUASH Score and Individual Physical Activity Categories' SQUASH Scores) Influenced by Occupation
Description: as for outcome 1
Time Frame: Month 0 and Month 12 LOCF
Population: Analysis included all participants who received at least one dose of adalimumab with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 381
units on a scale
  SQUASH (Manual job, N=184) | 1235.3 (4853.6)
  SQUASH (Non-manual job, N=189) | 518.4 (4160.2)
  SQUASH-A (Manual job, N=188) | 62.2 (977.3)
  SQUASH-A (Non-manual job, N=193) | -131.3 (1100.4)
  SQUASH-B (Manual job, N=185) | 614.5 (3452.2)
  SQUASH-B (Non-manual job, N=189) | 544.1 (2799.3)
  SQUASH-C (Manual job, N=186) | 456.6 (1875.8)
  SQUASH-C (Non-manual job, N=192) | -53.0 (1535.6)
  SQUASH-D (Manual job, N=188) | 40.1 (1486.4)
  SQUASH-D (Non-manual job, N=193) | 151.7 (1590.1)

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the time the participant's informed consent was received until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment i.e., up to 12 months.
Description: Non serious adverse events were not collected for this study.
Arm/Group | Participants With Rheumatoid Arthritis
Serious Adverse Events (participants affected / at risk) | 32/460
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Rheumatoid Arthritis (N=460)
LEUKOPENIA (Blood and lymphatic system disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
CARDIAC FAILURE (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
CHEST PAIN (General disorders) | 1
NO THERAPEUTIC RESPONSE (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 2
BRONCHITIS (Infections and infestations) | 1
CYTOMEGALOVIRUS HEPATITIS (Infections and infestations) | 1
HERPES OPHTHALMIC (Infections and infestations) | 1
LOCALISED INFECTION (Infections and infestations) | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 1
TONSILLITIS (Infections and infestations) | 1
VAGINAL INFECTION (Infections and infestations) | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
LUPUS-LIKE SYNDROME (Musculoskeletal and connective tissue disorders) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
INTERCOSTAL NEURALGIA (Nervous system disorders) | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2
PHOTODERMATOSIS (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.